CLINICAL TRIAL: NCT01223690
Title: A Double-blind Randomized Placebo-controlled Clinical Trial of the Safety and Efficacy of Intravenous Clarithromycin as Immunomodulatory Therapy for the Management of Sepsis
Brief Title: Clarithromycin as Immunomodulator for the Management of Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Evangelos Giamarellos-Bourboulis, Assistant Professor of Medicine, Evangelos Giamarellos-Bourboulis, Assistant Professor of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A06-269
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2010-10

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: sepsis; infection; bacteremia; clarithromycin
MeSH Terms: conditions — Sepsis; Shock, Septic; Infections; Bacteremia | interventions — Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 250 ml of dextrose 5% administered intravenously within one hour of continuous infusion for four consecutive days
  Interventions: Drug: Dextrose 5%
- Clarithromycin (Active Comparator): 1000 mg of clarithromycin diluted in 250 ml of dextrose 5% administered intravenously within one hour of continuous infusion for four consecutive days
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin — 1000 mg diluted into 250 ml of dextrose 5% administered intravenously within one hour of continuous infusion for four consecutive days
  Other Names: Klaricid IV
  Arms: Clarithromycin
Drug: Dextrose 5% — 1000 mg diluted into 250 ml of dextrose 5% administered intravenously within one hour of continuous infusion for four consecutive days
  Other Names: Dextrose solution
  Arms: Placebo

SUMMARY:
The herein protocol is based on the results of one former clinical trial conducted by our study group showing the considerable efficacy of intravenously administered clarithromycin as an adjuvant to antimicrobial chemotherapy for patients with sepsis, septic shock and respiratory failure in the field of ventilator-associated pneumonia. The proposed clinical trial is based on the need to generalize the application of intravenous clarithromycin in the total of admitted septic patients irrespective of the underlying cause of sepsis.

DETAILED DESCRIPTION:
The idea for the application of intravenous clarithromycin as immunomodulatory therapy for the management of sepsis has been evolved on in vitro results showing that concentrations close to 10μg/ml may refrain biosynthesis of pro-inflammatory cytokines by inhibiting the activation of the translation factor NF-κB. Intravenously administered clarithromycin has been widely applied in experimental sepsis by one susceptible isolate of Escherichia coli, one multidrug-resistant isolate of Pseudomonas aeruginosa and one pan-resistant isolate of Klebsiella pneumoniae after induction of pyelonephritis by the test isolates. Results of these animal studies revealed that clarithromycin inhibited the evolution of the systemic inflammatory response syndrome (SIRS) acting at the cellular level of blood monocytes and that its effect was expressed when administered after induction of sepsis.

Based on the latter experimental data, one double-blind randomized clinical trail was conducted over the period June 2004-December 2005 in the 4th Department of Internal Medicine, in the 1st Department of Critical Care and in the 2nd Department of Critical Care of the University of Athens. The study enrolled 200 subjects with ventilator-associated pneumonia (VAP) and sepsis, severe sepsis or septic shock; 100 received placebo and 100 clarithromycin. Statistical analysis of results revealed that clarithromycin effected earlier resolution of signs of sepsis and of VAP accompanied by a) prolongation of survival of the total of patients over the first 16 days of follow-up, b) prolongation of survival of patients with septic shock for 28 days of follow-up, and c) 2.75-fold reduction of the relative risk of death over the first 28 days of follow-up in patients with multiple organ failure.

The proposed clinical trial is based on the extremely beneficial results of clarithromycin in the septic population of patients with VAP creating the following needs: a) to generalize the application of intravenous clarithromycin in the total of admitted septic patients irrespective of the underlying cause of sepsis, and b) to expand the effect of clarithromycin over a greater time period than the first 19 days post start of administration.

ELIGIBILITY:
Inclusion Criteria:

* One or more of the following infections: a) primary or secondary bacteremia by Gram-negative bacteria, b) acute pyelonephritis, or c) intrabdominal infection. Only one episode of infection per patient will be enrolled. Both patients with community-acquired and nosocomial infections are eligible for the study.
* The presence of at least two of the following criteria of sepsis according to ACCP/SCCM (8) a) body temperature >38 degreesC or <36 degreesC; b) pulse rate >90/min; c) breath rate >20/min or Pco2<32mmHg; and/or d) leukocytosis (white blood cell count >12,000/μl) or leukopenia (white blood cell count <4,000/μl) or >10% band forms

Exclusion Criteria:

* Presence of HIV infection
* Intake of corticosteroids at a dose more than or equal to 1mg/kg of equivalent prednisone for more than one month
* Neutropenia as <500 neutrophils/μl
* Selection by the attending physician of a macrolide as empiric antimicrobial therapy for the infection making the patient eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2007-07; Primary Completion 2010-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Effect of clarithromycin in mortality and risk for death by severe sepsis/shock and multiple organ dysfunction compared with placebo | 28 days
  Survival analysis for 28 days will be done between placebo-treated patients and clarithromycin-treated patients separately for patients with sepsis; for patients with severe sepsis; and for patients with septic shock. Odds ratios for death by septic shock and/or multiple organ dysfunction will be assessed separately for each arm. Comparison of odds ratios will be done.

SECONDARY OUTCOMES:
Effect of clarithromycin compared with placebo in time to resolution of infection | 28 days
  Time analysis between placebo-treated patients and clarithromycin-treated patients will be done
Effect of clarithromycin compared with placebo in time to resolution of sepsis | 28 days
  Time analysis between placebo-treated patients and clarithromycin-treated patients will be done
Effect of clarithromycin compared with placebo in time to progression to severe sepsis or septic shock and multiple organ failure | 28 days
  Time analysis between placebo-treated patients and clarithromycin-treated patients will be done
Influence of administration of clarithromycin compared with placebo on systemic inflammatory response | 10 days
  Comparative analysis of serum markers estimated at consecutive time intervals over the first 10 days of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, MD, PhD, Study Chair — National and Kapodistrian University of Athens; Helen Giamarellou, MD, PhD, Principal Investigator — National and Kapodistrian University of Athens; Apostolos Armaganidis, MD, Principal Investigator — National and Kapodistrian University of Athens; George Koratzanis, MD, Principal Investigator — Sismanogleion Athens General Hospital; Charalambos Gogos, MD, PhD, Principal Investigator — University of Patras; Konstantinos Atmatzidis, MD, Principal Investigator — University of Thessaloniki; Emmanouel Douzinas, MD, PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (6):
- Greece (6):
  - 3rd Department of Critical Care Medicine, National and Kapodistrian University of Athens, Athens
  - 2nd Department of Critical Care Medicine, National and Kapodistrian University of Athens, Athens
  - 4th Department of Internal Medicine, National and Kapodistrian University of Athens, Athens
  - 2nd Department of Medicine, Sismanogleion General Hospital, Athens
  - 1st Department of Medicine, University of Patras, Pátrai
  - 2nd Department of Surgery, University of Thessaloniki, Thessaloniki

REFERENCES:
- [Background] Giamarellos-Bourboulis EJ. Macrocycle molecules for the management of systemic infections: the clarithromycin paradigm. Curr Top Med Chem. 2010;10(14):1470-5. doi: 10.2174/156802610792232033. PMID 20536418
- [Background] Giamarellos-Bourboulis EJ, Pechere JC, Routsi C, Plachouras D, Kollias S, Raftogiannis M, Zervakis D, Baziaka F, Koronaios A, Antonopoulou A, Markaki V, Koutoukas P, Papadomichelakis E, Tsaganos T, Armaganidis A, Koussoulas V, Kotanidou A, Roussos C, Giamarellou H. Effect of clarithromycin in patients with sepsis and ventilator-associated pneumonia. Clin Infect Dis. 2008 Apr 15;46(8):1157-64. doi: 10.1086/529439. PMID 18444850
- [Background] Giamarellos-Bourboulis EJ, Tziortzioti V, Koutoukas P, Baziaka F, Raftogiannis M, Antonopoulou A, Adamis T, Sabracos L, Giamarellou H. Clarithromycin is an effective immunomodulator in experimental pyelonephritis caused by pan-resistant Klebsiella pneumoniae. J Antimicrob Chemother. 2006 May;57(5):937-44. doi: 10.1093/jac/dkl084. Epub 2006 Mar 20. PMID 16549515
- [Background] Giamarellos-Bourboulis EJ, Adamis T, Laoutaris G, Sabracos L, Koussoulas V, Mouktaroudi M, Perrea D, Karayannacos PE, Giamarellou H. Immunomodulatory clarithromycin treatment of experimental sepsis and acute pyelonephritis caused by multidrug-resistant Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2004 Jan;48(1):93-9. doi: 10.1128/AAC.48.1.93-99.2004. PMID 14693524
- [Derived] Vittoros V, Kyriazopoulou E, Lada M, Tsangaris I, Koutelidakis IM, Giamarellos-Bourboulis EJ. Soluble fms-like tyrosine kinase 1, placental growth factor and procalcitonin as biomarkers of gram-negative sepsis: Analysis through a derivation and a validation cohort. Medicine (Baltimore). 2021 Nov 5;100(44):e27662. doi: 10.1097/MD.0000000000027662. PMID 34871241
- [Derived] Karakike E, Kyriazopoulou E, Tsangaris I, Routsi C, Vincent JL, Giamarellos-Bourboulis EJ. The early change of SOFA score as a prognostic marker of 28-day sepsis mortality: analysis through a derivation and a validation cohort. Crit Care. 2019 Nov 29;23(1):387. doi: 10.1186/s13054-019-2665-5. PMID 31783881
- [Derived] Gainaru G, Papadopoulos A, Tsangaris I, Lada M, Giamarellos-Bourboulis EJ, Pistiki A. Increases in inflammatory and CD14dim/CD16pos/CD45pos patrolling monocytes in sepsis: correlation with final outcome. Crit Care. 2018 Mar 3;22(1):56. doi: 10.1186/s13054-018-1977-1. PMID 29499723
- [Derived] Antonakos N, Tsaganos T, Oberle V, Tsangaris I, Lada M, Pistiki A, Machairas N, Souli M, Bauer M, Giamarellos-Bourboulis EJ. Decreased cytokine production by mononuclear cells after severe gram-negative infections: early clinical signs and association with final outcome. Crit Care. 2017 Mar 9;21(1):48. doi: 10.1186/s13054-017-1625-1. PMID 28274246